CLINICAL TRIAL: NCT05502523
Title: The Impact of Surgical Technique on Circulating Tumor DNA in Early-Stage Non-Small Cell Lung Cancer
Brief Title: The Impact of Surgical Technique on Circulating Tumor DNA in Stage I-III Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22D.435; JT 19625 (Other: JeffTrial Number)
Record Dates: First submitted 2022-08-01; First posted 2022-08-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage I Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (pulmonary vein first approach procedure) (Active Comparator): Patients undergo pulmonary vein first approach surgical procedure on day of surgery.
  Interventions: Procedure: Pulmonary Artery-First Surgical Technique
- Group II (pulmonary artery first surgical procedure) (Active Comparator): Patients undergo pulmonary artery first approach surgical procedure on day of surgery.
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Pulmonary Artery-First Surgical Technique — Undergo pulmonary artery first surgical technique
  Other Names: Artery-First Technique; A-First Technique; Lung Cancer Artery-First Surgical Technique; Artery-First Surgical Technique; Artery-First Ligation
  Arms: Group I (pulmonary vein first approach procedure)
Procedure: Biospecimen Collection — Correlative studies
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Group II (pulmonary artery first surgical procedure)

SUMMARY:
This clinical trial compares the effect of pulmonary vein-first surgical technique to pulmonary artery-first surgical technique in decreasing circulating tumor cell deoxyribonucleic acid (ctDNA) in patients with stage I-III non-small cell lung cancer. Pulmonary vein first and pulmonary artery first surgical techniques are standard surgical techniques for the division of the blood vessels during lung resection surgery. Pulmonary vein-first surgical technique may reduce the risk of shedding tumor cells during surgery and influence long term overall survival.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the association between sequence of surgical resection and postoperative ctDNA levels at specified time points.

SECONDARY OBJECTIVE:

I. To determine the associated between sequence of surgical resection and postoperative ctDNA level and clinical oncologic outcomes.

II. To assess disease-free survival and the role of circulating tumor DNA in disease recurrence in patients with resectable non-small cell lung cancer.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients undergo pulmonary vein first approach surgical procedure on day of surgery.

GROUP II: Patients undergo pulmonary artery first approach surgical procedure on day of surgery.

After completion of surgery, patients are followed up at day 1, day 7, days 7-28, 4 months, every 6 months for 2 years, then every 6 months for up to 5 years

ELIGIBILITY:
Inclusion Criteria:

* Any patients 18 years of age or older with confirmed or suspected early-stage (stage I-III) NSCLC
* Eligible and scheduled for surgical anatomic lung resection (e.g. lobectomy or segmentectomy) as routine clinical care for their disease

Exclusion Criteria:

* Previous cancer diagnosis within 5 years (except ductal carcinoma in situ [DCIS] of the breast, superficial bladder cancer, non-melanoma skin primary, other malignancy that does not require treatment).
* Preoperative chemotherapy, immunotherapy, or radiation therapy
* Receipt of perioperative blood transfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Circulating tumor deoxyribonucleic acid (ctDNA) status | At postoperative day 2
  Stratified by surgical vascular division technique. A peripheral blood sample will be taken at the time of surgery to determine baseline ctDNA status. Following surgical resection a blood sample will be taken at specified time points (postoperative day 2; postoperative day 14) to determine ctDNA levels compared to baseline. The difference in the proportion of patients who have positive ctDNA status between those undergoing division/ligation in a "pulmonary-vein first" technique compared to a "pulmonary-artery first" technique will be estimated. The risk difference will be estimated along with a 95% confidence interval.
Circulating tumor deoxyribonucleic acid (ctDNA) status | At postoperative day 14
  Stratified by surgical vascular division technique. A peripheral blood sample will be taken at the time of surgery to determine baseline ctDNA status. Following surgical resection a blood sample will be taken at specified time points (postoperative day 2; postoperative day 14) to determine ctDNA levels compared to baseline. The difference in the proportion of patients who have positive ctDNA status between those undergoing division/ligation in a "pulmonary-vein first" technique compared to a "pulmonary-artery first" technique will be estimated. The risk difference will be estimated along with a 95% confidence interval.

SECONDARY OUTCOMES:
Disease free survival rate | Up to 5 years
  The distribution of survival outcomes will be estimated using the Kaplan-Meier method, stratified by ctDNA status at 2 days and 2 weeks. Key statistics (median survival, 1- and 2-year survival) will be estimated from the curve along with 95% confidence intervals. We will also use a Cox proportional hazard regression model, stratified by stage in the analyses, to estimate the hazard ratio along with a 95% confidence interval.
Overall survival rate | Up to 5 years
  The distribution of survival outcomes will be estimated using the Kaplan-Meier method, stratified by ctDNA status at 2 days and 2 weeks. Key statistics (median survival, 1- and 2-year survival) will be estimated from the curve along with 95% confidence intervals. We will also use a Cox proportional hazard regression model, stratified by stage in the analyses, to estimate the hazard ratio along with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Grenda, MD, Principal Investigator — TJU
Locations (4):
- United States (4):
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Jefferson Health Northeast, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Asplundh Cancer Pavilion at Jefferson Health, Willow Grove, Pennsylvania